CLINICAL TRIAL: NCT01514032
Title: TOP-Stone: Treatment of Patients With Small Kidney Stones - Randomized Head-to-head Trial Comparing Extracorporal Shockwave Lithotripsy With Retrograde Intrarenal Surgery
Brief Title: Extracorporal Shockwave Lithotripsy Versus Retrograde Intrarenal Surgery for the Treatment of Kidney Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOP-Stone
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi

ARMS (2):
- Extracorporal shockwave lithotripsy (Active Comparator)
  Interventions: Procedure: Extracorporal shockwave lithotripsy
- Retrograde intrarenal surgery (Active Comparator)
  Interventions: Procedure: Retrograde intrarenal surgery

INTERVENTIONS:
Procedure: Extracorporal shockwave lithotripsy — Extracorporal shockwave lithotripsy
  Arms: Extracorporal shockwave lithotripsy
Procedure: Retrograde intrarenal surgery — Retrograde intrarenal surgery
  Arms: Retrograde intrarenal surgery

SUMMARY:
The purpose of this study is to compare two established modalities for the treatment of kidneystones: ESWL (extracorporal shockwave-lithotripsy) vs. URS (uretero-reno-scopy with stone-extraction). Comparison of the stone-free rates 3month postoperative.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria: - kidneystones requiring treatment up to an maximal size of 15mm (singular or multiple kidneystones with at least one stone with min. 5mm of size)

* male and female patients between 18 and 99 years
* informed consent signed by patient after explanation of the both treatment-modalities

Exclusion criteria: - age < 18 or > 99

* pregnancy
* breastfeeding mother
* disorders of blood clotting
* kidneystones > 15mm
* aneurysms of the aorta or renal artery
* severe skeletal deformations which hamper one of the treatment modalities
* synchronous stones of the ipsilateral ureter
* stones which can not visualized which X-ray or sonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
stonefree-rates 3month after therapy | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Michael Muentener, MD, Principal Investigator — University Hospital Zurich, Division of urology
Locations (1):
- University Hospital Zurich, Urology, Zurich, Switzerland